CLINICAL TRIAL: NCT04872920
Title: Prospective, Multi-country, Observational Registry to Collect Clinical Information on Patients With Endogenous Cushing's Syndrome to Assess Drug Utilization Pattern and to Document the Safety and Effectiveness of Ketoconazole.
Brief Title: Observational Registry on Patients With Endogenous CS to Document Safety and Effectiveness of Ketoconazole.
Acronym: KetoPASS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: HRA Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: Keto PASS
Record Dates: First submitted 2021-02-16; First posted 2021-05-05 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Cushing Syndrome
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional, prospective, multinational, multicentre, observational study, in which data collected are those derived from routine clinical practice via an European registry on CS: ERCUSYN.

DETAILED DESCRIPTION:
The aim is to further document the safety and efficacy of Ketoconazole HRA administered in routine clinical practice in patients with CS.

The study operates under real clinical practice conditions, i.e. there is no treatment protocol thus.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged from 12 years or older with a diagnosis of CS
2. Patients who started ketoconazole therapy after study start
3. For patients previously treated with ketoconazole, patients must have taken their last dose at least 6 months before starting ketoconazole again in this study.
4. Written informed consent signed prior to registration of any patient data in HRA modules.

Exclusion Criteria:

1. Adrenal cortical carcinoma
2. Patients currently participating in any other trial (interventional or not) of an investigational medicine or participation in the past one month before start of ketoconazole
3. Patients who have at least one contraindication among those listed in section 4.3 of the ketoconazole SmPC

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include all patients aged 12 years and above with endogenous CS from all causes exposed to ketoconazole and included by the participating centers in ERCUSYN. Patients with CS due to an adrenal carcinoma will be excluded from the study population since adrenal carcinoma is excluded from ERCUSYN registry.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
incidence of hepatotoxicity and QT prolongation to assess liver and cardiac tolerability profile of ketoconazole. | up to 5 years of follow up
  The primary objective is to document liver and cardiac tolerability profile of ketoconazole p.o when administered as monotherapy or in combination with other therapies, in routine clinical practice, in patients with CS.

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 5 years of follow up
  Number of adverse events with Ketoconazole in monotherapy or in combination with other therapies for Cushing Syndrome.
Drug utilization pattern regarding safe utilization of ketoconazole according to HRA SmPC recommendations on liver function | up to 5 years of follow up
  Number of liver tests performed per patient Number of patients for whom LFTs were performed according to SmPC recommendations.
  Number of patients with reduction of ketoconazole dose following liver enzymes increase Number of patients with interruptions / definitive stop of ketoconazole following liver enzymes increase
Drug utilization pattern of ketoconazole according to HRA SmPC recommendations on liver function | up to 5 years of follow up
  Timing of liver tests performed per patient according to defined windows.
Drug utilization pattern regarding safe use of ketoconazole according to HRA SmPC recommendations on liver function | up to 5 years of follow up
  Percentage of patients for whom LFTs were performed according to SmPC recommendations.
  Percentage of patients with reduction of ketoconazole dose following liver enzymes increase Percentage of patients with interruptions / definitive stop of ketoconazole following liver enzymes increase
Drug utilization pattern regarding safe utilization of ketoconazole according to HRA SmPC recommendations on Qt interval monitoring. | up to 5 years of follow up
  Number of ECGs performed per patient Number of patients for whom ECGs were performed according to SmPC recommendations
Drug utilization pattern of ketoconazole according to HRA SmPC recommendations on Qt interval monitoring. | up to 5 years of follow up
  Timing of ECGs performed per patient according to defined windows
Drug utilization pattern regarding safe use of ketoconazole according to HRA SmPC recommendations on Qt interval monitoring. | up to 5 years of follow up
  Percentage of patients for whom ECGs were performed according to SmPC recommendations
Effectiveness of ketoconazole | up to 5 years of follow up
  clinical outcome evaluated by the physician after ketoconazole treatment: cortisol levels improvement or normalization after ketoconazole treatment clinical symptoms of Cushing Syndrome over time. Number and type of comorbidities. Number of concomitant treatments for comorbidities by drug class.
Impact on Quality of life, European Quality of Life questionnaire | up to 5 years of follow up
  self-administered questionnaire of Health-Related Quality of Life to evaluate current health regarding mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and the perceived health status of the patient.
  The answers given can be converted into utility scores anchored at 0 for death and 1 for perfect health. The questionnaire also includes a Vi-sual Analog Scale (VAS), by which respondents can reporttheir perceived health status with a grade ranging from 0(the worst possible health status) to 100 (the best possiblehealth status).
Impact on Quality of life, Cushing Quality of Life questionnaire | up to 5 years of follow up
  items referring to problems relevant to patients with CS with five categories of response.
  Answers are rated on a scale of 1-5, where '1' corresponds to 'Always' or 'Very much' and '5' to 'Never' or 'Not at all'. Therefore, the lower the score, the greater the impact on Health-Related Quality of Life.

CONTACTS AND LOCATIONS:
Locations (6):
- University Hospital Zagreb, Zagreb, Croatia
- France (3):
  - Hôpital Universitaire Grenoble, Grenoble
  - Hôpital Bicêtre APHP, Le Kremlin-Bicêtre
  - Hôpital de la Conception, Marseille
- Institut de Recerca de la Santa Creu i Sant Pau, Barcelona, Spain
- Sahlgrenska University Hospital, Gothenburg, Sweden